CLINICAL TRIAL: NCT05199766
Title: HEMolyse and Organ Damage imPROvement in Sickle Cell Disease by VoxElotor. An Open-label One Stage Phase II Design
Brief Title: Hemolysis Related Complications in SCD. A Phase II Study With Voxelotor
Acronym: HEMOPROVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP200750; 2020-005424-11 (EudraCT Number)
Record Dates: First submitted 2021-12-06; First posted 2022-01-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Hemolysis; Plasma Hemoglobin
MeSH Terms: conditions — Anemia, Sickle Cell; Hemolysis | interventions — voxelotor; WW Domain-Containing Oxidoreductase; Hemoglobin, Sickle

STUDY DESIGN:
Intervention Model Description: This is an open-label, single-arm, single-stage phase II trial in patients treated with Voxelotor 1500 mg daily for 48 weeks.
  Assessments will be done during the study at week 0, week 6, week 12, week 24, week 36 and week 48.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Voxelotor 1500 mg oral per day (GBT440) for 48 weeks (Experimental): Voxelotor 1500 mg oral per day (GBT440) for 48 weeks, in case of discontinuation due to patient's wishes and/or adverse event above grade 2 : 1000mg during 14 days then complete discontinuation if no resolution. In case of sudden discontinuation a therapeutic phlebotomy will be authorized.
  Interventions: Drug: Voxelotor 1500 mg oral per day (GBT440) for 48 weeks in patients with sickle-cell disease

INTERVENTIONS:
Drug: Voxelotor 1500 mg oral per day (GBT440) for 48 weeks in patients with sickle-cell disease — This is an open-label, single-arm, single-stage phase II trial of voxelotor in patients with sickle-cell disease. Voxelotor 500mg tablets. Voxelotor will be administered as 500mg tablets orally once daily. The participant should always take all 3 tablets in a row at the same time each day, unless the study doctor has instructed them to adjust the dose.

SUMMARY:
Intro:

Sickle cell disease is a genetic disorder caused by a mutation of the β hemoglobin called HbS, which causes red blood cell (RBC) abnormalities responsible for hemolysis, mainly intravascular, leading to chronic anemia. Intravascular hemolysis is responsible for severe inflammation and endothelial dysfunction.

Maintaining hemoglobin in its oxygenated R-conformation is one of the strategies for inhibiting the polymerization of HbS. Previous experimental therapeutic approaches having this effect have been discontinued due to poor pharmaceutical properties or toxicity. Nevertheless, they proved the validity of the concept by demonstrating an increase in oxyhemoglobin and a decrease in biomarkers of hemolysis.

Voxelotor binds to the α chain of globin and maintains Hb in its R conformation, thereby inhibiting the polymerization of HbS while increasing the affinity of Hb for oxygen.

Because of its mechanism of action affecting anemia and hemolysis, Voxelotor is a promising treatment for the prevention and treatment of renal and cerebral arterial disease.

Hypothesis/Objective :

Investigator hypothesis is that the treatment by Voxelotor (GBT440) will improve intra vascular hemolysis and will increase the total mass of hemoglobin with beneficial effects on organ function.

The primary objective of the study is to evaluate the biological activity of Voxelotor on the reduction of intra vascular hemolysis measured by plasma hemoglobin.

The secondary objectives of the study will aim at characterizing the effects of GBT 440 Voxelotor on:

* Intra vascular hemolysis measured by plasma Heme
* Total hemoglobin mass (MHb)
* RBCs lifespan
* Blood volumes (plasma volume (PV), red blood cell mass (RBCM), total blood volume (BV))
* Blood viscosity
* Cerebral perfusion
* Cerebrovascular vaso-reactivity
* Cognitive function (MoCA)
* Six minute walk test
* Renal perfusion and iron deposits in renal cortex
* Measurement of Glomerular filtration rate Estimation of glomerular filtration rate (CKD/EPI equation)
* Urine albumin/creatinine ratio
* Ability to decrease or stop erythropoietin in patients under EPO treatment
* Safety (VOC, ACS, Priapism) and tolerability of voxelotor
* RBC properties

Method:

This is an open-label, single-arm, single-stage phase II trial in patients treated with Voxelotor 1500 mg daily for 48 weeks. Assessments will be done during the study at week 0, week 6, week 12, week 24, week 36 and week 48.

ELIGIBILITY:
Inclusion Criteria:

* SS or S-β0 major sickle cell syndrome
* Hemoglobin level < 9 g/dL
* Aged 18 years or older
* Stable dose for at least 3 months if treated with HU, EPO, angiotensin-converting enzyme (ACE) or inhibitor/angiotensin receptor blocker (ARB) therapy; at least after 6 months after initiating HU treatment
* Patient with social security
* Female patient must have a negative serum pregnancy test (betaHCGat inclusion W0-V1D1) or evidence of post-menopausal status
* Effective methods of birth control (e.g., condom, spermicidal gel, oral contraceptive, indwelling intrauterine device, hormonal implant/patch, injections, approved cervical ring) or abstinence from screening through 4 weeks after last Voxelotor dose.

Exclusion Criteria:

-If patient does not have any of the following treatments (HU, Crizanlizumab) he will then be excluded if: Patient meets, at screening, Hydroxyurea/ Crizanlizumab indications of treatment (recurrent painful vaso-occlusive crises, including acute chest syndrome), even if these treatments are inappropriate (e.g. hematologic toxicity antecedent) or if the patient refuses these treatments

* Patients in chronic transfusion program or transfused < 3 months before enrolment
* Patient with severe organ involvement: hepatic (TP <50%), renal (eGFR<30 ml / ml/1.73m2 according to CKD/EPI or cardiac (LVEF <45%)
* Transplant patients.
* Pregnancy.
* Breast feeding patients
* Homeless patient
* Patient deprived of liberty by judicial or administrative decision or patient under guardianship
* Patient unable to understand the purpose and conditions of the study and unable to give consent
* Chronic use of NSAIDs (more than 10 days by month)
* Auto immune disease or infection not controlled or cancer
* VIH, HBV, HCV current infection
* Prior drug hypersensitivity to Voxelotor or excipients
* Known allergy or hypersensitivity to imaging contrast product
* Ongoing therapeutic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-03-22 (Estimated); Study Completion 2025-03-22 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the biological activity of voxelotor on the change of intra vascular hemolysis measured by decrease of plasma hemoglobin. | Change from Baseline at Week 48
  Change of Intravascular hemolysis, as defined by a ≥20% decrease of plasma Hemoglobin (µmol/l)

SECONDARY OUTCOMES:
Intra vascular hemolysis measured by plasma Heme | Week 0, Week 24, Week 48
  Absolute and relative (%) changes in plasma Hemoglobin (µmol/l) and free plasma Heme (µmol/l)
Total hemoglobin mass (MHb) | Week 0, Week 24, Week 48
  Measurement of total hemoglobin mass based on the CO rebreathing technique (g of Hb / kg), or a stable evolution (i.e. decrease ≤ 10%) in patients initially under EPO therapy and who decreased or discontinued EPO during the study period.
RBCs lifespan | Week 0, Week 24, Week 48
  RBC lifespan by measurement of alveolar CO (in days).
Change of blood volumes (plasma volume (PV) and total blood volume (BV)) | Week 0, Week 24, Week 48
  Blood volumes by CO rebreathing method (Total blood volume (L), Plasma Volume (L) )
Change of red blood cell mass (RBCM) | Week 0, Week 24, Week 48
  RBC mass (g)
Change of Total Mass of Hemoglobin | Week 0, Week 24, Week 48
  Total Mass of Hemoglobin (g of Hb)
Change of blood viscosity | Week 0, Week 24, Week 48
  Blood viscosity (cP)
Cerebral perfusion | Week 0, Week 24, Week 48
  Cerebral perfusion measured by MRI
Change of cerebrovascular vaso-reactivity measured by transcranial Doppler | Week 0, Week 24, Week 48
  Transcranial Doppler (Breath holding test)
Change of cerebrovascular vaso-reactivity measured by Near Infra Red Spectroscopy | Week 0, Week 24, Week 48
  Cerebral vaso-reactivity measured by Near Infra Red Spectroscopy
Cognitive function (MoCA) | Week 0, Week 24, Week 48
  Cognitive performance measured by MoCA Improvement in the 6 minutes walk test on : Time spent under Sp02 88 and 90%, Borg Rating of Perceived Exertion (RPE), distance.
Measurement of renal perfusion and amount of deoxyhemoglobin | Week 0, Week 24, Week 48
  Amount of deoxyhemoglobin by MRI
Study of iron deposits in renal cortex | Week 0, Week 24, Week 48
  Iron deposits in renal cortex measured by MRI
Measurement of Glomerular filtration rate | Week 0, Week 24, Week 48
  Estimation of glomerular filtration rate (CKD/EPI equation)
Ability to decrease or stop erythropoietin in patients under EPO treatment | From Week 0 to Week48
  Concomitant treatment observation: decrease / interruption of EPO dose
Incidence of Treatment-Adverse Events VOC, ACS and Priapism | From Week 0 to Week48
  Presence/Absence of adverse Events VOC, ACS, Priapism

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Andre Natella, PHD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
APHP IS DATA'S OWNER, PLEASE CONTACT BOARD

REFERENCES:
- [Derived] Liu W, Kassasseya C, Papamanolis L, Nguyen-Peyre KA, Garreau M, Eckert S, De Luna G, d'Humieres T, de Pierrefeu V, Arnaud C, Bekeziz N, Metteil MPG, Provost C, Gerbeau JF, Verlhac S, Bartolucci P, Vignon-Clementel I. Vascular Geometry Drives Stroke Risk in Sickle Cell Disease. Am J Hematol. 2026 Jan 28. doi: 10.1002/ajh.70184. Online ahead of print. PMID 41603130